CLINICAL TRIAL: NCT05717322
Title: The Effect of Transcutaneous Stimulation (TENS) on the Recovery of Muscle Function After Orthognathic Surgery
Brief Title: TENS and Orthognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, lecturer of oral and maxillofacial surgery, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC2227
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Orthognathic Surgery
Keywords: orthognathic; TENS; EMG
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS arm (Experimental)
  Interventions: Behavioral: TENS
- non TENS arm (Active Comparator)
  Interventions: Behavioral: sham TENS

INTERVENTIONS:
Behavioral: TENS — apply TENS after orthognathic surgery
  Arms: TENS arm
Behavioral: sham TENS — apply non active TENS after orthognathic surgery
  Arms: non TENS arm

SUMMARY:
All patients with skeletal deformity will undergo orthognathic surgery after orthodontic treatment. After surgery TENS electrodes( rubber electrodes with the same size 5.3×4.8 cm) will be Placed bilaterally on ant temporalis and bilaterally on superficial masseter muscle…Time : 30 min /3 times per week/ 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Class II facial deformity
* absence of temporomandibular joint pain and preoperative opening mouth limitation
* normal cranial form
* presence of dentition
* Fit to GA

Exclusion Criteria:

* temporomandibular joint pain and preoperative opening mouth limitation;
* craniofacial anomalies and abnormal cranial form
* absence of facial trauma, mandibular condylar fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-01-22 (Actual); Primary Completion 2024-01-22 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
maximum mouth opening | 6 months
  will be measured by
  caliber between the incisal edges of upper and lower centrals

SECONDARY OUTCOMES:
visual analogue scale | 6months
  will be measured by VAS scale at the same time points of mouth opening(0_10) 0 represent no pain,10represent high pain
muscle activity | 6months
  measured by EMG at the same time points

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt